CLINICAL TRIAL: NCT05091190
Title: Immunotherapy Clearance and Phenotype of Circulating Tumor Cells in Patients With Lung and Head and Neck Cancers, Treated With an Immunotherapy-based Therapy
Brief Title: Immunotherapy Clearance and Phenotype of Circulating Tumor Cells in Lung and Head and Neck Cancers
Acronym: MADMAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_0458; 2021-A01482-39 (Other: ID-RCB)
Record Dates: First submitted 2021-09-01; First posted 2021-10-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Metastatic NSCLC; Metastatic Head and Neck Cancer
Keywords: metastatic NSCLC; metastatic head and neck cancer; clearance; PD-L1; CTCs; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cancer patients (Other): MADMAS will include 30 patients with metastatic NSCLC and 30 patients with metastatic head and neck cancers; patients will NSCLC will receive an immunotherapy-based treatment in first line metastatic setting; patients with head and neck cancers are included if they are planned to receive an immunotherapy-based treatment, whatever the line.
  Interventions: Other: Blood draws

INTERVENTIONS:
Other: Blood draws — Blood draws will be realized at the following time points:
  C1T1: at the baseline, before treatment administration. C1T2: cycle 1, after treatment administration. C2T1: the day of the 2nd cycle, before treatment administration. C2T2: the day of 2nd cycle, after treatment administration. C3T1: the day of the 3rd cycle, before treatment administration. C3T2: the day of 3rd cycle, after treatment administration.

SUMMARY:
Immunotherapy is widely administrated as anticancer treatment in metastatic setting. Despite a proved efficacy in several cancer types and clinical situations, it exists a wide variability of responses in terms of efficacy and toxicity. The rate of responders depends mostly on the type of pathology, with 40% of responders among melanoma patients, 20-30% among lung and head and neck cancer patients and only 1% of responders among pancreatic cancer patients. Thus, the main challenge today is to be able to select patients for whom the treatment is likely to be effective. Several studies suggested that tumors with a high mutational burden and expressing PD-L1 are better responders to immunotherapy.

However, a proportion of PD-L1 negative cancers responds to immunotherapy, suggesting that other parameters have to be considered together with PD-L1 expression. Of that, the immunotherapy clearance seems to have an impact on overall survival, but larger studies, including different molecules and cancer types, are needed to better understand the correlation between the clearance and the response to immunotherapy.

Tumor cells released from the primary tumor in the blood circulation (CTCs, for circulating tumor cells) are considered as "liquid biopsies", as they contain the entire genetic and phenotypic information representative of the tumor, including PD-L1 expression. Thus, the variation of PD-L1 expression under treatment can be easily followed-up on blood samples collected during the time.

The objective of MADMAS is to study the correlation between the immunotherapy clearance, measured at the different times during treatment, and the variation of the number of CTCs expressing PD-L1 after two cures of treatment.

MADMAS will enroll patients with lung or head and neck cancers, treated with an immunotherapy-based therapy. Blood samples will be collected at the baseline and before the first two cures of treatment. The immunotherapy clearance will be measured with an innovative approach of Mass Spectrometry, and PD-L1 expression will be measured on CTCs, purified with a highly sensitive microfluidics technology.

ELIGIBILITY:
Inclusion Criteria:

Lung cancer (n= 30):

* Adult patients
* Patients who gave its written informed consent to participate to the study
* Weight at inclusion ≥ 48 kg
* NSCLC histology only
* Stage IV according to 8th TNM classification
* Planned to be treated with immunotherapy (+/- chemotherapy) as a first line treatment in metastatic setting
* PD-L1 status on primary tumor available at the inclusion
* Patients affiliated to a social insurance regime

Head and neck cancer (n= 30):

* Adult patients
* Patients who gave its written informed consent to participate to the study
* Weight at inclusion ≥ 48 kg
* Recurrent or metastatic epidermoid carcinomas from oral cavity, oropharynx, hypopharynx, larynx (except nasopharynx)
* Stage IV according to 8th TNM classification
* Planned to be treated with immunotherapy (+/- chemotherapy)
* PD-L1 status on primary tumor available at the inclusion
* Patients affiliated to a social insurance regime

Exclusion Criteria:

* History of previous cancers, except for adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, treated and with no evidence of disease for ≥ 5 years
* Patients under tutorship or guardianship
* Pregnant or breast feeding women
* Patients under psychiatric care

Exclusion Criteria specific pour head and neck cohort:

- Patients already treated with immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Immunotherapy clearance (mL/min) and number of PD-L1 (absolute number) positive CTCs after two cycles of treatment (composite criteria) | At the end of cycle 2 (each cycle is 21 days)
  The clearance and the number of PD-L1 positive cells will be measured on blood samples collected the day of the third immunotherapy administration (each cycle is 14 to 28 days, depending on the type of immunotherapy).

SECONDARY OUTCOMES:
Overall survival | 2 years
  time elapsed between the first immunotherapy administration and the death
Progression free survival | 2 years
  time elapsed between the first immunotherapy administration and progression
level of PD-L1 expression on primary tumor tissue | 2 years
  The level of PD-L1 expression will be measured by ICH on tissue from primary tumor surgery/biopsy through study completion, an average of 2 years.
Baseline transcriptomic profile of CTCs isolated form peripheral blood | Day 1 of cycle 1, before treatment administration (cycle length: 14 days for nivolumab treatment and 21 days for pembrolizumab treatment)
  Baseline transcriptomic profile of CTCs isolated form peripheral blood: the transcriptomic profile of CTCs will be analyzed by NGS (Next-Generation Sequencing) from blood samples collected at cycle 1 day 1, before treatment administration.
1st cycle transcriptomic profile of CTCs isolated form peripheral blood | Day 1 of cycle 2, before treatment administration (cycle length: 14 days for nivolumab treatment and 21 days for pembrolizumab treatment)
  The transcriptomic profile of CTCs will be analyzed by NGS (Next-Generation Sequencing) from blood samples collected after the 1st cycle of treatment (cycle length between 14 and 21 days depending on the type of immunotherapy)
2nd cycle transcriptomic profile of CTCs isolated form peripheral blood | Day 1 of cycle 3, before treatment administration (cycle length: 14 days for nivolumab treatment and 21 days for pembrolizumab treatment)
  The transcriptomic profile of CTCs will be analyzed by NGS (Next-Generation Sequencing) from blood samples collected at the end of cycle 2 (each cycle is 21 days).
identification of CTCs transcriptomic signatures, associated to immunotherapy efficacy or toxicity | 2 years
  the CTCs transcriptomic profile (measure 4) will be obtained with the NGS method; the analyses of these profiles will imply statistical models of logistic regression (Lasso Method). These data will be compared with clinical data on efficacy (PFS measured at 2 years after the beginning of treatment) and toxicity (stopping treatment for toxicity before the third cycle).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PHILOUZE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Croix Rousse Hospital, Lyon
  - Lyon Sud Hospital, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No